CLINICAL TRIAL: NCT04384237
Title: Effect of Er,Cr: YSGG Laser - Aided Circumferential Supracrestal Fiberotomy in the Prevention of the Lower Incisors Rotational Relapse
Brief Title: Er,Cr:YSGG Laser-aided Fiberotomy in the Prevention of the Lower Incisors Rotational Relapse
Acronym: laser
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación Universitaria CIEO (Other)
Responsible Party: Principal Investigator, Sandra Leal, Docent, Fundación Universitaria CIEO
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CIEO
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Rotated Teeth
Keywords: Conventional supracrestal Fiberotomy; Laser -aided Fiberotomy; Er;Cr:YSGG Laser; Incisors rotation relapse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (outcomes Assessor) An external clinic is going to do the measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Er,Cr:YSGG laser-aided CSF (Experimental): Experimental: Er, Cr: YSGG laser-aided Circumferential Supracrestal Fiberotomy in the lower arch, posterior leveling and alignment of the orthodontic treatment by inserting the laser tip at an angle of 10-15º to the radicular surface
  Interventions: Procedure: Er,Cr:YSGG laser-aided CSF
- Conventional CSF (Active Comparator): Fiberotomy comparator: this arm is going to receive a blade conventional Circumferential Supracrestal Fiberotomy in the lower arch, posterior leveling and alignment by inserting a surgical blade into the gingival sulcus at an angle like that in the laser-aided CSF.
  Interventions: Procedure: Conventional CSF

INTERVENTIONS:
Procedure: Er,Cr:YSGG laser-aided CSF — After injection 2% lidocaine with 1:80.000 epinephrine concentration in labial and lingual vestibule the fiberotomy is carried out by inserting a 9 x 0.5 mm laser tip into the gingival sulcus with an angle of 10-15º to the radicular surface
  Arms: Er,Cr:YSGG laser-aided CSF
Procedure: Conventional CSF — After injection 2% lidocaine with 1:80.000 epinephrine concentration in labial and lingual vestibule the fiberotomy is carried out by inserting a surgical blade (#11)into the gingival sulcus at an angle of 10-15º to the radicular surface
  Arms: Conventional CSF

SUMMARY:
To establish the effect of erbium, chromium,yttrium,scandium,gallium and garnet (Er,Cr: YSGG) laser-aided circumferential supracrestal fiberotomy compared to a conventional circumferential supracrestal fiberotomy group, after leveling and alignment during the first month after arch wire removal on the prevention of rotational relapse in lower incisors.

Methods: Randomized clinical trial in 60 orthodontic patients with two to four lower incisors rotation between 30º-50º degrees before treatment.They are going to be assigned in two intervention groups, each group with 30 patients. One group are going to be treated with Er;Cr: YSGG laser -aided CSF and the other group with conventional circumferential supracrestal fiberotomy. After leveling and alignment each procedure will be performed and after one month healing the arch wire will be removed for a month and lower incisor relapse will be measured through cast models in a software. Periodontal parameters will be registered before and after procedures.The outcomes are going to be determined and compared between groups with corresponding statistical test and results will be analyzed

DETAILED DESCRIPTION:
(Population, intervention, comparison, outcomes )PICO QUESTION Is there any difference in the amount of rotational relapse of the anterior lower teeth after leveling and alignment between Er;Cr:YSGG laser-aided circumferential supracrestal fiberotomy compared with conventional circumferential supracrestal fiberotomy after the removal of the arch wire one month once healed?

Population: Orthodontic patients with lower incisors rotation between 30º-50º degrees

Intervention:Er:Cr;YSGG Laser-aided CSF (Waterlase, Biolase, Irvine,California, USA) Comparison: Conventional CSF

Outcomes Primary Outcome: rotation relapse degree after one month removed teeth from the arch wire Secondary Outcome: probing depth and clinical crown height (gingival margin position)baseline, after leveling and alignment stage one month removed lower incisors from the arch wire.

AIMS

GENERAL AIM

To establish the effect of Er,Cr: YSGG laser -aided circumferential supracrestal fiberotomy compared to a conventional circumferential supracrestal fiberotomy group on the prevention of rotational relapse in lower incisors, during the first month after the teeth are removed from the arch.

SPECIFIC AIMS

* Determine the degree of rotation of the lower incisors in the two groups of the pretreatment study, at the end of the alignment and leveling stage and the month after performing the intervention.
* Determine the probing depth and the position of the gingival margin of the lower incisors in the two groups of the pretreatment study, at the end of the alignment and leveling stage and the month after performing the intervention.
* Determine the perception of pain in patients of the two study groups at baseline, 24, 48 and 72 hours.
* Compare rotational relapse, probing depth, gingival margin position in each study group during the follow-up time.
* Compare rotational relapse, probing depth and gingival margin position between study groups during follow-up time.

METHODS

OVERVIEW OF DESIGN Study design: Randomized clinical trial

Randomized clinical trial in 60 lower incisors with moderate initial rotation (30-50 degrees). The eligible patients are going to be randomly allocated into two groups, each group with 30 teeth.

One group is going to be treated with Er,Cr:YSGG laser - aided circumferential supracrestal fiberotomy and the other group with conventional circumferential supracrestal fiberotomy.

Blinding: it is not possible to blind patients and clinical staff, but the investigators are going to blind the operator who will perform the measurements and the data analysis (single-blinded)

The protocol for both procedures will be the same except for the intervention.

Alginate impressions and cast models at the beginning of the study will be taken and initial rotation of mandibular incisors will be measured based on a Xerox copy of the lower cast (Canon Xerox Machine, imageRUNNER (IR) 5050 Ota, Tokyo, Japan) while the occlusal table faced down on the screen, a Xerox copy of it will be made. The Xerox copies will be scanned (Canon CanoScan 9000F Mark II, Ota, Tokyo, Japan) and saved as a image file format JPEG (Joint Photographic Experts Group) files. The files will be imported to the software to drawn an imaginary arch passing through the outermost surface of the anterior and posterior teeth.

To measure the initial rotation, the JPEG images will be opened in a Digimizer image analysis software (Version 4.3 Orange, California)The angle between the incisor edge and the line tangent to the imaginary arch will be measured as initial rotation.

Measures of lower incisors will be taken by previously-calibrated operators as well as periodontal measurements at baseline, after leveling and alignment and one month after separating the teeth from the arch wire.

Pain measurement evaluations will be determined by the visual analogue scale (VAS) at baseline, 24,48 y 72 hrs.

DESIGN FOR SAMPLING

Study Population:

-Orthodontic patients from the orthodontic department clinics of the UniCieo

Sampling:

No probabilistic: convenience sample Consecutive sample of consenting patients

PLANS FOR RECRUITMENT

Patients of the Clinic University (UniCieo) that meet the selection criteria and accept to participate.

MEASUREMENTS

MAIN PREDICTOR VARIABLE

-Relapse lower incisors (Er;Cr YSGG laser-aided CSF)

POTENTIAL CONFOUNDING

Age

Sex

OUTCOME VARIABLES

Dental stone cast scanned Outcomes (T3-T4):

-Quantity of lower anterior teeth rotation relapse tendency measured 1 month after arch wire removed

Periodontal Outcomes:

Quantity of probing depth and gingival margin position (coronal height) measured 1 month after arch wire removed

Pain Outcomes:

Visual analogue scale (0-10) measures after clinical intervention

STATISTICAL ISSUES

APPROACH TO STATISTICAL ANALYSIS

The data analysis will be processed in the statistics program Statistical Package for the Social Sciences (SPSS) software (version 21, Chicago, IL).Evaluation of normality of data will be valued with the Kolmogorov-Smirnov test. One-way ANOVA will be used to determine any significant differences Significance level is going to be set at P< 0.05

ELIGIBILITY:
Inclusion Criteria:

* Non gingivitis or untreated caries
* lower teeth with 30º-50º rotation degree
* 2 mm keratinized tissue band
* at least 2 rotated mandibular teeth

Exclusion Criteria:

* Root canal treatment
* Marginal Recessions
* Interproximal bone loss in Rx
* Thin gingival biotype (periodontal probe translucency
* Reduced periodontium
* systemic diseases or medications that alters bone metabolism.
* Pregnancy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Quantity of anterior mandibular rotation relapse | one month after arch wire removal
  Er,Cr.YSGG laser-aided fiberotomy and Conventional CSF. Alginate impressions and cast models at the beginning of the study.Herb curve to measure the initial rotation grade. Impressions and measurements after the leveling and alignment phase, fiberotomy procedure, retention for one healing month. 30 days later of the removal of the arch wire, alginate impressions and measures will be taken by previously-calibrated operators

SECONDARY OUTCOMES:
Changes in probing depth | baseline and two months after fiberotomy
  At the beginning of the study, two months after fiberotomy, measures will be taken by calibrated operators
Changes in clinical crown height | baseline and two months after fiberotomy
  At the beginning of the study, two months after fiberotomy, measures will be taken by calibrated operators
Pain levels | after procedures, 24, 48 and 72 hours
  Pain levels will be measure by the Visual Analog Scale (VAS), from 0 to 10-cm VAS, where the number 0 indicating no pain, a value less than 4 on the EVA means mild pain, between 4 and 6 moderate pain, greater than 6 very intense pain and the number 10 indicating the most severe pain into the scale, after 24, 48 and 72 hours CSF procedures

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Plaza, Ms., Study Director — Fundación Universitaria CIEO
Locations (1):
- Orthodontic Clinic of Post-graduation Program UniCIEO, Bogotá, Bogota D.C., Colombia